CLINICAL TRIAL: NCT03074474
Title: A Prospective, Single Arm, Multi-center Study Evaluating the Short-term Clinical Outcomes of Ventral Hernias Treated With OviTex Reinforced Bioscaffold.
Brief Title: Ventral Hernia Study Using OviTex Reinforced Bioscaffold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tela Bio Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TB2016.01.01
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Hernia, Ventral
Keywords: use of mesh
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- OviTex Permanent 1S (Other): All subjects included in this post-market study had a ventral hernia repaired with OviTex 1S Permanent reinforced tissue matrix.
  Interventions: Device: OviTex 1S Permanent

INTERVENTIONS:
Device: OviTex 1S Permanent — OviTex 1S Permanent is a reinforced tissue matrix consisting of layers of extra-cellular matrix derived from sheep stomachs. The layers are embroidered together with a monofilament polypropylene. One side of the mesh has blue polypropylene stitching, which provides a surface conducive to native tissue growth. The other side of the mesh is a smooth surface intended to minimize tissue attachment (adhesions).

SUMMARY:
The study is designed to demonstrate that the use of OviTex® 1S material for a ventral hernia repair leads to the same or a lower percentage of early post-operative complications and true hernia recurrences when compared to other types of available meshes. 100 subjects will be included from 5-7 participating investigator sites. Within 30 days prior to the hernia repair surgery, a baseline visit will be performed during which the patient's eligibility for the study will be evaluated. The surgical technique used for the repair will be determined by the investigator/surgeon. Additional study data will be collected during the hospital stay, 30 and 90 days post-operatively and 12 and 24 months post-operatively. At the follow up visits, the surgical site will be evaluated by the surgeon, both the surgeon and patient will be asked to rate their satisfaction with the repair and the subject will be asked to complete two Quality of Life questionnaires.

DETAILED DESCRIPTION:
The study is intended to evaluate the post-operative complications and re-herniations following the use of OviTex® Permanent 1S reinforced bioscaffold in subjects with ventral hernias. The study is designed to mirror surgical standard of care for ventral hernia intervention, with the exception of asking for subjects to return for evaluation at longer time points post-surgery than is typical for standard care. A baseline visit will be performed for patients who are identified for and provide informed consent to participate in the study. During this visit, a review of medical history, a physical exam and assessment of the hernia site will be performed. The potential subject will also be asked to complete two quality of life surveys; one that is disease specific and one that is a standard method of health assessment. On the day of surgery, the ventral hernia will be repaired with the use of OviTex® 1S reinforced bioscaffold. Perioperative data will be collected and the surgeon will provide an assessment of the product's handling qualities. During the course of the hospital stay, the subject will be assessed for incidence of early post-operative surgical site wound events and complications, all necessary medical interventions and/or re-operations. On the day of discharge, surgical site occurrences or wound related events noted at the hernia repair site and the occurrence of other post-operative complications will be assessed.

The Day 30 and Day 90 visits will have a visit window of +/- 2 weeks. At these visits, the incidence of late surgical site occurrences or wound related events noted at the hernia repair site will be assessed. If hernia recurrence is suspected, it will be confirmed via diagnostic imaging with a CT scan. The occurrence of other late post-operative complications will also be assessed. The subjects will be asked to complete the same disease specific questionnaire and the same health assessment questionnaire as was done at the Baseline visit, however the subject will also be asked to complete a pain assessment. Both the surgeon and the subject will provide an assessment of his/her satisfaction with the hernia repair. The activities at Months 12 and 24 mirror those of Days 30 and 90, however the visit window is extended to +/- 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject suffers from an uncomplicated ventral hernia that requires surgical repair (open, laparoscopic, or robotic) with the use of an implant to reinforce or replace weakened or missing tissue.
* The size of the implant needed for repair is expected to be 18 x 22 cm, 20 x 20 cm or less.
* Subject meets CDC/SSI Wound Classification Class I (Clean), Class II (Clean-Contaminated) or Class III (Contaminated) criteria
* Subject is willing and able to sign an informed consent for the study and has signed the IRB approved Informed Consent form for this study.
* Subject is able to complete Quality of Life (QoL) and pain Questionnaires.
* Subject is at least 18 years old (or considered an adult per state law).
* Subject is able to participate fully in, and for the full duration of, the study.

Exclusion Criteria:

* Subject has a BMI of > 40.
* Subject meets CDC/SSI Wound Classification Class IV(Dirty-Infected) criteria.
* Subject is female and is pregnant.
* Subject has a life expectancy of < 2 years making it unlikely that the subject will successfully achieve two-year follow-up.
* Subject has recent history of drug or alcohol abuse (in last 3 years).
* Subject has an allergy to ovine-derived products.
* Subject has participated in another clinical trial within the past 30 days or is currently involved in another clinical trial.
* Subject is unable to receive OviTex® Permanent 1S reinforced bioscaffold at the time of surgery.

Intra-operative Exclusion Criteria

* Subject requires implant that exceeds 18 x 22 cm or 20 x 20 cm.
* Subject unable to receive OviTex® Permanent 1S reinforced bioscaffold at time of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2021-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George DeNoto, MD, Principal Investigator — Saint Francis Hospital
Locations (7):
- United States (7):
  - Scripps Clinic, La Jolla, California
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - St. Luke's Hospital South, Overland Park, Kansas
  - Capital Health, Trenton, New Jersey
  - St. Francis Hosptial, Roslyn, New York
  - Comanche County Memorial Hospital, Lawton, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] DeNoto G 3rd, Ceppa EP, Pacella SJ, Sawyer M, Slayden G, Takata M, Tuma G, Yunis J. 24-Month results of the BRAVO study: A prospective, multi-center study evaluating the clinical outcomes of a ventral hernia cohort treated with OviTex(R) 1S permanent reinforced tissue matrix. Ann Med Surg (Lond). 2022 Sep 27;83:104745. doi: 10.1016/j.amsu.2022.104745. eCollection 2022 Nov. PMID 36389188
- [Derived] DeNoto G 3rd, Ceppa EP, Pacella SJ, Sawyer M, Slayden G, Takata M, Tuma G, Yunis J. A Prospective, Single Arm, Multi-Center Study Evaluating the Clinical Outcomes of Ventral Hernias Treated with OviTex(R) 1S Permanent Reinforced Tissue Matrix: The BRAVO Study 12-Month Analysis. J Clin Med. 2021 Oct 27;10(21):4998. doi: 10.3390/jcm10214998. PMID 34768516

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 95 patients were consented, 3 did not meet eligibility criteria and were not enrolled. Only 92 patients were enrolled in the study and received OviTex 1S Permanent reinforced tissue matrix during their hernia repair procedure.
Period: Overall Study
Arm/Group | OviTex Permanent 1S
Started | 92
Completed | 65
Not Completed | 27
Not completed — Lost to Follow-up | 10
Not completed — Withdrawal by Subject | 10
Not completed — Death | 4
Not completed — 1 exited due to recurrence and 2 exited due to mesh removal. | 3

BASELINE CHARACTERISTICS:
Population: 95 subjects consented for participation in the study. 3 subjects did not meet all eligibility criteria and as such, 92 subjects were enrolled and underwent hernia repair procedures with OviTex 1S.
Arm/Group | OviTex Permanent 1S
Number analyzed (Participants) | 92
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 60.42 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 91
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 88
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: (kg/m^2)] | 31 (4.51)
modified Ventral Hernia Working Group Grade [Count of Participants; unit: Participants] — Modified Ventral Hernia Working Group Grade is used to predict surgical site occurrence (SSO) based on patient comorbidities. Grade I patients are considered to have a low risk of complications and have no history of wound infection. Grade 2 patients are considered a higher risk for developing an SSO and have one of the following comorbidities: diabetes, COPD, immunosuppression, active smoker, or obese. Grade 3 patients are at the highest risk for developing an SSO and are considered contaminated with a stoma present, violation of gastrointestinal tract, infected mesh, or septic dehiscence
  Participants
    Grade I | 21
    Grade II | 52
    Grade III | 19
Surgical Site Wound Classification [Count of Participants; unit: Participants]
  CDC Class I Clean | 74
  CDC Class II Clean-Contaminated | 14
  CDC Class III Contaminated | 4
Operative Approach [Count of Participants; unit: Participants]
  Open | 60
  Laparoscopic | 12
  Robotic | 20
Plane of Placement [Count of Participants; unit: Participants]
  Retrorectus/TAR | 48
  Intraperitoneal | 42
  Retrofascial/Pre-Periotneal | 1
  Onlay | 1

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Occurrences or Wound-related Events
Description: The primary endpoints were number of participants experiencing an SSO or wound related event at the hernia repair site and the number of participants experiencing other complications <90 days after index surgery. These included seromas, hematomas, wound dehiscence, skin necrosis, fistulae, and infections. Complications such as ileus and bowel obstruction were also recorded.
Time Frame: within the first three months of the ventral hernia repair
Measure: Count of Participants; unit: Participants
Groups:
- OviTex 1S Permanent: All subjects included in this post-market study had a ventral hernia repaired with OviTex 1S Permanent reinforced tissue matrix.
Arm/Group | OviTex 1S Permanent
Number analyzed (Participants) | 92
Participants
  Adjacent Recurrence | 0
  Seroma | 10
  Seroma (requiring intervention) | 3
  Hematoma | 4
  Wound Dehiscence | 1
  Skin Necrosis | 1
  Fistulae | 2
  Surgical Site Infection | 15
  Bowel Obstruction | 1
  Ileus | 8
  Any other non-surgery or hernia-related complications | 1
  Mesh Removal (Full) | 1
  Mesh Removal (Partial) | 1
  Superficial Infection | 9
  Deep/Abscess Infection | 6
  Organ Space Infection | 0

2. Secondary Outcome: Hernia Recurrence, Post-operative SSO, and Wound Related Events at the Hernia Repair Site Occurring at Time Points > 90 Days After Index Surgery
Description: Secondary outcome measures include the number of participants experiencing a hernia recurrence, post-operative SSO, wound related event at the hernia repair site, and other complications occurring at time points > 90 days after index surgery.
Time Frame: Overall Cumulative SSOs and Complications (0 - 24 Months)
Measure: Count of Participants; unit: Participants
Arm/Group | OviTex 1S Permanent
Number analyzed (Participants) | 92
Participants
  Adjacent Recurrence | 3
  Seroma | 12
  Seroma (requiring intervention) | 3
  Hematoma | 4
  Wound Dehiscence | 1
  Skin Necrosis | 1
  Fistulae | 2
  SSI | 19
  Bowel Obstruction | 1
  Ileus | 8
  Any other non-surgery or hernia-related complication | 2
  Mesh removal (full) | 2
  Mesh removal (partial) | 1

3. Secondary Outcome: Change in Patient Reported Outcomes (HerQLes) From Baseline to Each Time Point
Description: Hernia-Related Quality-of-Life Survey (HerQLes) assesses abdominal wall function and impact of ventral hernia repair on quality of life through 12 questions. Responses are graded on a likert scale from 1 to 6, 1=strongly disagree, 2=moderately disagree, 3=slightly disagree, 4=slightly agree, 5=moderately agree, 6=strongly agree. A raw score is calculated by the following formula:
  12 question average = (Response to Q1 + Response to Q2 +…+ Response to Q12) / 12
  A summary score is calculated by the following formula:
  HerQLes Summary Score = 120-20*(12 Question Average) HerQLes scores range from 0 (worst possible response) to 100 (best possible response).
  Data is reported as change in HerQLes Summary Score from baseline to each time point The scale was first reported in Krpata, D. M. et al. Design and Initial Implementation of HerQLes: A Hernia-Related Quality-of-Life Survey to Assess Abdominal Wall Function. J Am Coll Surgeons 215, 635-642 (2012).
Time Frame: Baseline through 24 months
Population: The number of participants at each time point differs from the overall number of participants analyzed (92) as not all participants completed the required questionnaires at each time point and therefore, only the questionnaires that were available to be analyzed are included.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OviTex 1S Permanent
Number analyzed (Participants) | 92
scores on a scale
  Day 30: number analyzed (Participants) | 81
  Day 30 | -5.67 (31.62)
  Day 90: number analyzed (Participants) | 76
  Day 90 | 16.25 (31.12)
  Month 12: number analyzed (Participants) | 70
  Month 12 | 25.03 (30.09)
  Month 24: number analyzed (Participants) | 59
  Month 24 | 26.93 (29.01)

4. Secondary Outcome: Change in Patient Reported Outcomes (EQ-5D VAS) From Baseline to Each Time Point
Description: EuroQol 5 Dimensions (EQ-5D) Visual Analog Scale (VAS) is a standardized generic (disease non-specific) quality of life scale measuring how good or bad the patients' health is on their visit date. The patient indicates on the scale from 0 (the worst health you can imagine) to 100 (the best health you can imagine) how their health is with an X and reports the number in a box.
  Data is reported as change in EQ-5D VAS score from baseline to each time point.
Time Frame: Baseline through 24 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OviTex 1S Permanent
Number analyzed (Participants) | 92
scores on a scale
  Day 30: number analyzed (Participants) | 82
  Day 30 | -0.05 (19.49)
  Day 90: number analyzed (Participants) | 77
  Day 90 | 0.49 (21.21)
  Month 12: number analyzed (Participants) | 70
  Month 12 | 6.70 (20.48)
  Month 24: number analyzed (Participants) | 60
  Month 24 | 5.28 (18.97)

5. Secondary Outcome: Change in Patient Reported Outcomes (EQ-5D Index) From Baseline to Each Time Point
Description: EuroQol 5 Dimensions (EQ-5D) is a standardized generic (disease non-specific) quality of life instrument measuring mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Responses are coded from 1 to 5 (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, 5=extreme problems). The levels reported for each dimension create a 5-digit number (i.e. 11111 or 12345) based on patient response. These 5-digit numbers are converted to an index score by special algorithm that is not publicly available. The index value represents the patient's health status, where higher numbers are associated with better outcomes. Data is reported as change in EQ-5D Index value from baseline to each time point.
Time Frame: Baseline through 24 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OviTex Permanent 1S
Number analyzed (Participants) | 92
scores on a scale
  Day 30: number analyzed (Participants) | 81
  Day 30 | -0.048 (0.150)
  Day 90: number analyzed (Participants) | 77
  Day 90 | 0.006 (0.164)
  Month 12: number analyzed (Participants) | 70
  Month 12 | 0.046 (0.142)
  Month 24: number analyzed (Participants) | 60
  Month 24 | 0.042 (0.129)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from all study subjects from the time of the index surgery through the 24 month follow-up.
Groups:
- OviTex 1S Permanent: All subjects included in this post-market study will have a ventral hernia repaired with OviTex 1S Permanent reinforced tissue matrix.
Arm/Group | OviTex 1S Permanent
All-Cause Mortality (participants affected / at risk) | 4/92
Serious Adverse Events (participants affected / at risk) | 34/92
Other Adverse Events (participants affected / at risk) | 24/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OviTex 1S Permanent (N=92)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Fistula of small intestine (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 5 (6)
Incision site abscess (Infections and infestations) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1)
Complications of transplanted liver (Injury, poisoning and procedural complications) | 1 (1)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OviTex 1S Permanent (N=92)
Constipation (Gastrointestinal disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 6 (7)
Pyrexia (General disorders) | 5 (5)
Seroma (Injury, poisoning and procedural complications) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT03074474/Prot_SAP_002.pdf